CLINICAL TRIAL: NCT03199092
Title: Effectiveness of Intervention for Developmental Dyslexia: Rhythmic Reading Training Compared to 'Abilmente' Method
Brief Title: Rhythmic Reading Training Compared to 'Abilmente' Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Alice Cancer, PhD candidate, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRT-Abilmente
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Developmental Dyslexia
Keywords: Reading; Developmental Dyslexia; Music; Rhythm; Intervention
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RRT+sat (Experimental): RRT in combination with specific auditory training (sat) administered for a total of 20 hours over 10 weeks (60 minutes biweekly sessions).
  Interventions: Behavioral: RRT+sat
- Abilmente (Experimental): Abilmente method administered for a total of 10 hours over 5 weeks (60 minutes biweekly sessions).
  Interventions: Behavioral: Abilmente

INTERVENTIONS:
Behavioral: RRT+sat — RRT is a child-friendly computerized reading training program designed for Italian students with DD aged 8-14 yrs. The main feature of this intervention is the integration of a traditional remediation approach (sublexical treatment) with rhythm processing. Therefore, all reading exercises are characterized by a rhythmic accompaniment with gradually increasing speed. For this study, RRT was delivered in combination with a specific auditory training involving several music games specifically designed for improving auditory processing abilities typically compromised in children with DD.
  Arms: RRT+sat
Behavioral: Abilmente — 'Abilmente' method is an intervention for DD that comprises several validated treatments resulting in a proposal tailored to meet individual needs and features.
  Arms: Abilmente

SUMMARY:
The purpose of the present study is to compare the effectiveness of Rhythmic Reading Training (RRT), a computer-assisted intervention method that combines sublexical reading exercises with rhythm processing, and that of a multimodal intervention comprising different methodology, called 'Abilmente'. All interventions were delivered for a period ranging 1-2,5 months, in 60 minutes biweekly sessions.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with DD (ICD-10 code: F81.0) on the basis of standard inclusion and exclusion criteria (ICD-10: World Health Organization, 1992) and of the diagnosis procedure followed in the Italian practice

Exclusion Criteria:

* presence of comorbidity with other neuropsychiatric or psychopathological conditions (whereas comorbidity with other learning disabilities were allowed)
* exclusion criteria for the use of tDCS (e.g. epilepsy, pregnancy).

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Text reading accuracy expressed in number of errors change | 1 month
  Text reading accuracy expressed in number of errors The ability to read aloud a text was assessed using the Italian standardized test 'Prove di lettura MT', which provides speed and accuracy scores in reading aloud age-normed texts.
Text reading speed expressed in syllables per seconds change | 1 month
  The ability to read aloud a text was assessed using the Italian standardized test 'Prove di lettura MT', which provides speed and accuracy scores in reading aloud age-normed texts.
Word reading speed expressed in syllables per seconds change | 1 month
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Word reading accuracy expressed in number of errors change | 1 month
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Pseudo-word reading speed expressed in syllables per seconds change | 1 month
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).
Pseudo-word reading accuracy expressed in number of errors change | 1 month
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).
Text reading accuracy expressed in number of errors change | 2.5 months
  Text reading accuracy expressed in number of errors The ability to read aloud a text was assessed using the Italian standardized test 'Prove di lettura MT', which provides speed and accuracy scores in reading aloud age-normed texts.
Text reading speed expressed in syllables per seconds change | 2.5 months
  The ability to read aloud a text was assessed using the Italian standardized test 'Prove di lettura MT', which provides speed and accuracy scores in reading aloud age-normed texts.
Word reading speed expressed in syllables per seconds change | 2.5 months
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Word reading accuracy expressed in number of errors change | 2.5 months
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Pseudo-word reading speed expressed in syllables per seconds change | 2.5 months
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).
Pseudo-word reading accuracy expressed in number of errors change | 2.5 months
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Antonietti, PhD, Study Director — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - Catholic University of the Sacred Heart, Milan
  - Studio Abilmente, Milan